CLINICAL TRIAL: NCT06271785
Title: ISEPEE : Prognostic Value of High-resolution Electrical Source Imaging on the Success of Pediatric Focal Epilepsy Surgery
Brief Title: Prognostic Value of High-resolution Electrical Source Imaging on the Success of Pediatric Focal Epilepsy Surgery
Acronym: ISEPEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49RC22_0354
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HR-EEG recording (Experimental)
  Interventions: Diagnostic Test: HR-EEG recording

INTERVENTIONS:
Diagnostic Test: HR-EEG recording — All participants will have a HR-EEG recordings. It will be made at rest. Nap-like sleep is encouraged, but no sedatives will be given. Recording time will not exceed two hours.

SUMMARY:
This study investigates the usefulness of high resolution electrical source imaging (HR-ESI) in the setting of presurgical evaluation of drug-resistant focal epilepsy in children.

This method is based on an estimation of the intra-cerebral source that produces a signal recorded by scalp electrodes by solving the inverse problem, taking into account attenuation factors resulting from particular conductivity properties of the cerebral, peri-cerebral and cranial tissues.

Electrical sources are then fused on structural magnetic resonance imaging (MRI).

Scalp EEG recorded using 64 to 256 electrodes refers to as high resolution EEG (HR-EEG), leading to HR-ESI.

Studies based on small population of children or on mixt population of children and adults showed that HR-ESI has accuracy values, i.e. percentage of true positives (electrical source localized in the brain area resected and success of surgery) and true negatives (electrical source localized outside the brain area resected and failure of surgery) among the total population, ranging from 50 to 80%.

Discrepancies between studies could be explained by the limited number of patients included or by the mixture of pediatric and adult data.

Another limitation of previously published studies is that the spatial pattern of dipole source distribution was not taken into account to determine prediction accuracy of ESI.

Studies using magnetoencephalography (MEG) to perform magnetic source imaging (MSI) suggest that the spatial pattern of dipole source distribution needs to be considered, a spatially-restricted dipole distribution being associated with better post-surgical outcome when resected.

To tackle these issues, the investigators aim to conduct the first large prospective multicentric study in children with focal epilepsy candidates to surgery to assess prediction accuracy of ESI based on the finding of tight clusters of dipoles.

This is original as this pattern (tight versus loose cluster of dipoles) has been studied by several researchers using MEG but not using HR-EEG.

The investigators make the hypothesis that HR-EEG will allow to identity good candidates for epilepsy surgery and thus to offer this underutilized treatment in more children with better post-surgical outcome.

Among the secondary objectives, the investigators will address methodological issues related to the resolution of the inverse problem (methods using distributed sources models versus methods based on equivalent dipole estimation), the potential added value to model high-frequency oscillations (HFO), and the investigators will assess the cost-utility of the HR-ESI procedure.

DETAILED DESCRIPTION:
This study investigates the usefulness of high resolution electrical source imaging (HR-ESI) in the setting of presurgical evaluation of drug-resistant focal epilepsy in children.

This method is based on an estimation of the intra-cerebral source that produces a signal recorded by scalp electrodes by solving the inverse problem, taking into account attenuation factors resulting from particular conductivity properties of the cerebral, peri-cerebral and cranial tissues.

Electrical sources are then fused on structural magnetic resonance imaging (MRI).

Scalp EEG recorded using 64 to 256 electrodes refers to as high resolution EEG (HR-EEG), leading to HR-ESI.

Studies based on small population of children or on mixt population of children and adults showed that HR-ESI has accuracy values, i.e. percentage of true positives (electrical source localized in the brain area resected and success of surgery) and true negatives (electrical source localized outside the brain area resected and failure of surgery) among the total population, ranging from 50 to 80%.

Discrepancies between studies could be explained by the limited number of patients included or by the mixture of pediatric and adult data.

Another limitation of previously published studies is that the spatial pattern of dipole source distribution was not taken into account to determine prediction accuracy of ESI.

Studies using magnetoencephalography (MEG) to perform magnetic source imaging (MSI) suggest that the spatial pattern of dipole source distribution needs to be considered, a spatially-restricted dipole distribution being associated with better post-surgical outcome when resected.

To tackle these issues, the investigators aim to conduct the first large prospective multicentric study in children with focal epilepsy candidates to surgery to assess prediction accuracy of ESI based on the finding of tight clusters of dipoles.

This is original as this pattern (tight versus loose cluster of dipoles) has been studied by several researchers using MEG but not using HR-EEG.

The investigators make the hypothesis that HR-EEG will allow to identity good candidates for epilepsy surgery and thus to offer this underutilized treatment in more children with better post-surgical outcome.

Among the secondary objectives, the investigators will address methodological issues related to the resolution of the inverse problem (methods using distributed sources models versus methods based on equivalent dipole estimation), the potential added value to model high-frequency oscillations (HFO), and the investigators will assess the cost-utility of the HR-ESI procedure.

The study focuses on epileptic children who are candidates to a procedure of epilepsy surgery aiming to make them seizure-free. The principle of epilepsy surgery is to remove the brain area that generates patient's seizures, i.e. the seizure onset zone (SOZ). Candidates are patients with focal seizures that do not completely respond to the medical treatment and impact their quality of life. This represents 5-10% of epileptic children. Pre-surgical evaluation of these patients consists to perform in a first step non-invasive methods aimed to localize the SOZ: video-EEG in order to characterize usual seizures of the patient and to record and localize interictal epileptiform discharges (IED), MRI to search for a structural epileptogenic lesion, and positron emission tomography (PET) with fluorodeoxyglucose (FDG) to search for a brain area showing abnormal FDG uptake. After this so-called phase 1 work-up, the case is discussed in a multidisciplinary meeting, resulting in one of the 3 following decisions: (1) surgical resection when information from phase 1 is considered as sufficient, (2) continuation of the surgical process by performing a phase 2 evaluation, i.e. an invasive EEG recording using intracranial electrodes implanted by stereotaxy (SEEG), when information from phase 1 is considered as insufficient but made possible to pose a hypothesis regarding the localization of the SOZ, and (3) rejection for surgery. In children, epilepsy makes patient seizure-free in 60-80% of the cases. HR-ESI is a relatively new method that has been developed to localize non-invasively the SOZ with the hope to decrease the number of patients rejected for surgery or oriented to phase 2, and to increase the rate of success of epilepsy surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥2 and <17 years;
2. Drug-resistant focal epilepsy (failure of at least 2 well-conducted drug trials);
3. Phase 1 pre-op evaluation with scalp video-EEG recording, MRI and PET-FDG suggesting that the patient could be a good candidate for epilepsy surgery;
4. Recent scalp EEG record (within 12 months) showing the presence of interictal spikes;
5. High-quality and recent (within 6 months) structural MRI with 3D-T1 sequences covering the whole brain and the scalp available.

Exclusion Criteria:

1. Behavioral deficits making recording of scalp EEG impossible without sedation;
2. Informed consent form not signed by the parents;
3. Patient not affiliated to a social security system

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Prediction accuracy index | 24 months
  The main outcome is the prediction accuracy index, as assessed in fusing pre-op current equivalent dipoles to postop MRI, based on a tight cluster of spikes compared to the prediction accuracy index based on a loose cluster of spikes or on multiple clusters of spikes.

SECONDARY OUTCOMES:
Localization of the epileptogenic zone (Baseline) | Baseline
  To assess the ability of HR-ESI to localize the epileptogenic zone. Spatial congruence between the brain areas involved by the sources of interictal spikes and the epileptogenic zone, defined by either a MRI lesion concordant with the electroclinical data, or the brain area resected in patients who achieved good outcome following surgery.
Localization of the epileptogenic zone (After Surgery) | 24 months (= V3)
  To assess the ability of HR-ESI to localize the epileptogenic zone. Spatial congruence between the brain areas involved by the sources of interictal spikes and the epileptogenic zone, defined by either a MRI lesion concordant with the electroclinical data, or the brain area resected in patients who achieved good outcome following surgery.
preoperative accuracy of epileptogenic source localization | 12 months (= V2)
  To determine the preoperative accuracy of epileptogenic source localization delineated by HR-ESI.
  Spatial congruence between the brain areas involved by the sources of interictal spikes and the SOZ as assessed by intracranial EEG in patients oriented to intracranial EEG investigation.
prognostic value of HFO | 24 months (= V3)
  To determine the prognostic value of epileptogenic source localization delineated by HR-ESI based on high-frequency oscillations (HFO), on successful epilepsy surgery.
  Prediction accuracy index, as assessed in fusing pre-op current equivalent dipoles to postop MRI, based on of a unique, well delineated and completely resected cluster of HFO, compared to other situations.
Impact of method of sources reconstruction, conditions of EEG recordings and sampling rate | 3 months (= V1)
  To study the influence of some factors that could impact results of HR-ESI: type of method of sources reconstruction, conditions of EEG recordings (awake state versus sleep), and sampling rate.
  Congruence of the brain areas identified by HR-ESI according to the methods of sources reconstruction, the type of spikes (awake versus sleep) and the sampling rate.
health-economic modeling | 24 months (= V3)
  To perform a health-economic modeling to assess cost-utility and cost-effectiveness of the HR-ESI procedure. Evolution of Quality of life assessed with Child Health Utility 9 Dimensions (CHU9D) questionnaire

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Angers university hospital, Pédiatric department, Angers
  - Lille University Hospital, Clinical Neurophysiology Department, Lille
  - Civil Hospices of Lyon, Functional Neurology Department, Lyon
  - Marseille Timone University Hospital, Epileptology and Cerebral Rhythmology Department, Marseille
  - Nancy University Hospital, Neurology Department, Nancy
  - Paris Neck University Hospital, Pediatric department, Paris
  - Paris Robert-Debré University Hospital, Department of Physiology, Pediatric functional explorations, Paris
  - Rothschild Ophtalmologic Fondation, Pediatric neurosurgery Department, Paris
  - Rennes University Hospital, Pediatric department, Rennes

IPD SHARING:
Plan to Share IPD: No